CLINICAL TRIAL: NCT06707987
Title: An Open, Prospective, Non-interventional, Multicentre, Controlled Study of Safety and Efficacy of the Thrombolysis With the Non-immunogenic Staphylokinase in Patients With Acute Ischemic Stroke (FORPI Registry)
Brief Title: Post-registration Trial of the Non-immunogenic Staphylokinase in Acute Ischemic Stroke (FORPI Registry)
Status: Completed | Type: Observational
Sponsor: Supergene, LLC (Industry)
Collaborators: Federal Center of Cerebrovascular Pathology and Stroke, Russian Federation Ministry of Health (Other)
Responsible Party: Sponsor
Other Study IDs: FORPI
Record Dates: First submitted 2024-11-19; First posted 2024-11-27 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Fibrinolysis; Thrombolysis; Non-immunogenic staphylokinase
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-immunogenic staphylokinase: Drug: non-immunogenic staphylokinase
  Interventions: Drug: Non-immunogenic staphylokinase

INTERVENTIONS:
Drug: Non-immunogenic staphylokinase — Drug: non-immunogenic staphylokinase 10 mg as a single intravenous bolus Other Names: Fortelyzin®
  Other Names: Fortelyzin®

SUMMARY:
The aim of FORPI Registry is to study the safety and efficacy of the non-immunogenic staphylokinase in patients with acute ischemic stroke in routine clinical practice.

DETAILED DESCRIPTION:
Acute ischemic stroke is caused by the formation of blood clot in the major vessel which gives blood supply to a certain part of the brain. New approaches to the treatment of acute ischemic stroke include the use of modern highly effective methods of reperfusion of brain tissue in the first hours of the disease, aimed at restoring blood flow in the affected vessel, which helps prevent the development of irreversible damage to brain tissue or reduce its volume, i.e. minimize the severity of residual neurological deficit.

In December 2019, a multicenter, open-label, randomized non-inferiority trial of the efficacy and safety of the non-immunogenic staphylokinase (Fortelyzin®) compared with alteplase (Actilyse®) in patients with acute ischemic stroke (FRIDA) was completed (NCT03151993).

The primary efficacy outcome in both the non-immunogenic staphylokinase and alteplase groups, as well as in their subgroups depending on age, body weight, onset to treatment time, baseline NIHSS, localization and subtype of acute ischemic stroke showed that the non-immunogenic staphylokinase administered as a single bolus in a dose of 10 mg regardless of body weight is non-inferior to alteplase, administered as a bolus infusion at a dose of 0.9 mg/kg body weight, at a maximum dose of 90 mg in the treatment of patients with acute ischemic stroke within 4.5 hours from the symptoms onset. The non-immunogenic staphylokinase has demonstrated high safety profile. The indication "acute ischemic stroke" is included in the Instructions for medical use of the non-immunogenic staphylokinase. In routine clinical practice, the non-immunogenic staphylokinase is used for acute ischemic stroke treatment since 2021.

The aim of FORPI Registry is to study the safety and efficacy of the non-immunogenic staphylokinase in patients with acute ischemic stroke in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 years and older.
* Verified diagnosis of acute ischemic stroke.
* The time from the symptoms onset is no more than 4.5 hours.
* Thrombolysis with the non-immunogenic staphylokinase, 10 mg as a single intravenous bolus.

Exclusion Criteria:

* The time from the symptoms onset is more than 4.5 hours or the time of the symptoms onset is unknown.
* Increased sensitivity to the non-immunogenic staphylokinase.
* Systolic blood pressure above 185 mm Hg or diastolic blood pressure above 110 mm Hg or the need in the drug administration to reduce blood pressure to these levels.
* Neuroimaging (CT, MRI) signs of intracranial hemorrhage, brain tumors, arteriovenous malformation, brain abscess, aneurysm of cerebral vessels.
* Surgery on the brain or spinal cord.
* Suspicion of subarachnoid hemorrhage.
* Signs of severe stroke: clinical signs (stroke scale NIH > 25), neuroimaging (according to CT of the brain and / or MRI of the brain in the DWI, the ischemia focuses on the territory of more than 1/3 of the CMA pool).
* Simultaneous reception of oral anticoagulants, for example, warfarin with INR> 1.3.
* The use of direct anticoagulants (heparin, heparinoids) in the preceding stroke of 48 h with APTT values above the norm.
* Prior stroke or severe head injury within 3 months.
* Significant regression of neurological symptoms during the observation of the patient before thrombolysis.
* Hemorrhagic stroke or stroke, unspecified in history.
* Strokes of any genesis in the history of a patient with diabetes mellitus.
* Gastrointestinal bleeding or bleeding from the genitourinary system in the last 3 weeks. Confirmed exacerbations of gastric ulcer and duodenal ulcer during the last 3 months.
* Extensive bleeding now or within the previous 6 months.
* Severe liver disease, including liver failure, cirrhosis, portal hypertension (with varicose veins of the esophagus), active hepatitis.
* Acute pancreatitis.
* Bacterial endocarditis, pericarditis.
* Aneurysms of arteries, malformations of arteries and veins. Suspicion of exfoliating aortic aneurysm.
* Neoplasms with an increased risk of bleeding.
* Large operations or severe injuries within the last 14 days, minor surgery or invasive manipulation in the last 10 days.
* Puncture of uncompensated arteries and veins during the last 7 days.
* Prolonged or traumatic cardiopulmonary resuscitation (more than 2 min).
* Pregnancy, obstetrics, 10 days after birth.
* The number of platelets is less than 100,000 / μL.
* Blood glucose less than 2.7 mmol / L or more than 22.0 mmol / L.
* Hemorrhagic diathesis, including renal and hepatic insufficiency.
* Data on bleeding or acute trauma (fracture) at the time of examination.
* Seizures in the onset of the disease, if there is no certainty that the seizure is a clinical manifestation of acute ischemic stroke with a postictal residual deficiency.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 years and older with verified acute ischemic stroke, less than 4.5 h symptoms onset to treatment, who received a single intravenous bolus of the non-immunogenic staphylokinase (10 mg).
Sampling Method: Non-Probability Sample
Enrollment: 23250 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) score of 0-2 on day 90 after drug administration | day 90 after drug administration
  The number of patients with Modified Rankin Scale (mRS) scores 0-2 on day 90 after drug administration, where 0 - No symptoms, 1 - No significant disability, 2 - Slight disability.

SECONDARY OUTCOMES:
mRS score on day 90 after drug administration | day 90 after drug administration
  The median of mRS score on day 90 after drug administration, where:
  0 - No symptoms, 1 - No significant disability, 2 - Slight disability, 3 - Moderate disability, 4 - Moderately severe disability, 5 - Severe disability, 6 - Dead.
The National Institutes of Health Stroke Scale (NIHSS) at 24 hours after drug administration | 24 hours after drug administration
  The median of The National Institutes of Health Stroke Scale (NIHSS) at 24 h after drug administration, where: 0 - No stroke symptoms, 1-4 - Minor stroke, 5-15 - Moderate stroke, 16-20 - Moderate to severe stroke, 21-42 - Severe stroke.
NIHSS on day 7 after drug administration | day 7 after drug administration
  The median of NIHSS on discharge

OTHER OUTCOMES:
All-cause mortality | day 90 after drug administration
  The number of death from any causes during 90 days after drug administration
Intracranial haemorrhage | day 90 after drug administration
  The number of intracranial haemorrhage during 90 days after drug administration
Symptomatic intracerebral haemorrhage | day 90 after drug administration
  The number of symptomatic intracranial haemorrhage (sICH) defined as an NIHSS decline of ≥4 points compared with baseline NIHSS or the lowest NIHSS value or death between baseline and 7 days, associated with any haemorrhage judged by core lab evaluation to be responsible for the decline. Blood may be anywhere in the intracranial space including in the intraventricular, intraparenchymal and/or subarachnoid space (modified ECASS III definition) during 90 days after drug administration
Major bleedings | day 90 after drug administration
  The number of major bleedings (according to BARC classification type 3 and 5) during 90 days after drug administration
Thrombectomy | day 90 after drug administration
  The number of thrombectomy during 90 days after drug administration
Allergic reactions | day 90 after drug administration
  The number of allergic reactions during 90 days after drug administration
Pulmonary embolism | day 90 after drug administration
  The number of pulmonary embolism during 90 days after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay A. Shamalov, MD, PhD Prof, Principal Investigator — Federal Brain and Neurotechnology Center
Locations (1):
- Federal Brain and Neurotechnology Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gusev EI, Martynov MY, Nikonov AA, Shamalov NA, Semenov MP, Gerasimets EA, Yarovaya EB, Semenov AM, Archakov AI, Markin SS; FRIDA Study Group. Non-immunogenic recombinant staphylokinase versus alteplase for patients with acute ischaemic stroke 4.5 h after symptom onset in Russia (FRIDA): a randomised, open label, multicentre, parallel-group, non-inferiority trial. Lancet Neurol. 2021 Sep;20(9):721-728. doi: 10.1016/S1474-4422(21)00210-6. PMID 34418399
- [Background] Alasheev AM, Lantsova EV, Tretyakov DA. [Efficacy and safety of non-immunogenic staphylokinase in the ischemic stroke in real-world clinical practice in the Sverdlovsk region]. Zh Nevrol Psikhiatr Im S S Korsakova. 2023;123(7):74-79. doi: 10.17116/jnevro202312307174. Russian. PMID 37490668
- [Background] Ramazanov GR, Kokov LS, Shamalov NA, Kovaleva EA, Klychnikova EV, Akhmatkhanova LK, Cheboksarov DV, Khamidova LT, Muslimov RS, Rybalko NV, Petrikov SS. [First case of thrombolysis with non-immunogenic staphylokinase in a patient with ischemic stroke receiving dabigatran etexilate followed by thrombectomy]. Zh Nevrol Psikhiatr Im S S Korsakova. 2022;122(6):145-151. doi: 10.17116/jnevro2022122061145. Russian. PMID 35758961
- [Background] Kulesh AA, Syromyatnikova LI, Krapivin S, Astanin PV. [Comparison of the effectiveness of non-immunogenic staphylokinase and alteplase for intravenous thrombolysis in ischemic stroke: analysis of hospital registry data]. Zh Nevrol Psikhiatr Im S S Korsakova. 2024;124(7):139-144. doi: 10.17116/jnevro2024124071139. Russian. PMID 39113454
- [Background] Gusev EI, Martynov MY, Shamalov NA, Yarovaya EB, Semenov MP, Semenov AM, Orlovsky AA, Kutsenko VA, Nikonov AA, Aksentiev SB, Yunevich DS, Alasheev AM, Androfagina OV, Bobkov VV, Choroshavina KV, Gorbachev VI, Korobeynikov IV, Greshnova IV, Dobrovolskiy AV, Elemanov UA, Zhukovskaya NV, Zakharov SA, Chirkov AN, Korsunskaya LL, Nesterova VN, Nikonova AA, Nizov AA, Girivenko AI, Ponomarev EA, Popov DV, Pribylov SA, Semikhin AS, Timchenko LV, Jadan ON, Fedyanin SA, Chefranova ZY, Lykov YA, Chuprina SE, Vorobev AA, Archakov AI, Markin SS. [Nonimmunogenic staphylokinase in the treatment of acute ischemic stroke (FRIDA trial results)]. Zh Nevrol Psikhiatr Im S S Korsakova. 2022;122(7):56-65. doi: 10.17116/jnevro202212207156. Russian. PMID 35904293
- [Result] Shamalov NA, Martynov MY, Yarovaya EB, Chefranova ZY, Kutsenko VA, Semenov AM, Ivanov SV, Semenov MP, Markin SS, Gusev EI; FORPI Study Group. Thrombolysis With the Non-Immunogenic Staphylokinase for Acute Ischemic Stroke in the FORPI Registry: An Observational Study. Stroke. 2026 Feb;57(2):394-403. doi: 10.1161/STROKEAHA.125.051115. Epub 2025 Nov 26. PMID 41293810
- [Result] Shamalov NA, Chefranova ZY, Yarovaya EB, Kutsenko VA, Marskaya NA, Semenov AM, Semenov MP, Ivanov SV, Romashova YA, Markin SS. Prognostic outcome of intravenous thrombolysis with non-immunogenic staphylokinase in patients aged >/= 60 years with acute ischemic stroke by THRIVE scale. J Thromb Thrombolysis. 2025 Nov 16. doi: 10.1007/s11239-025-03212-0. Online ahead of print. PMID 41243072